CLINICAL TRIAL: NCT04798443
Title: Comparison of Subureteral Endoscopic Injection of Dextranomer/Hyaluronic Acid and Lich-Gregoir Ureteral Reimplantation In the Treatment of Pediatric Primary Vesicoureteral Reflux: Prospective Randomized Study
Brief Title: Endoscopic Injection of Dextranomer/Hyaluronic Acid Versus Ureteral Reimplantation In Treatment of Vesicoureteral Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsayed Salih (Other)
Responsible Party: Sponsor-Investigator, Elsayed Salih, assistant professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uro-surg./R/2015/0011
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Vesico-Ureteral Reflux
Keywords: Extravesical Reimplantation; Subureteral Injection; Vesico-ureteral reflux; Endoscopic; Dexell
MeSH Terms: conditions — Vesico-Ureteral Reflux | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subureteral endoscopic injection (Active Comparator): The endoscopic procedure was done under general anesthesia, and all patients received antibiotic prophylaxis. We used the subureteral injection technique (STING), as described by O'Donnell and Puri (1984). The volume of Dx/HA was injected until ureteral orifice collapse in all patients. The needle was held for 30 s.
  Interventions: Procedure: subureteral endoscopic Injection of Dextranomer/Hyaluronic acid (Dexell)
- open ureteral reimplantation (lich-gregoir) (Active Comparator): extravesical ureteral reimplantation (lich-gregoir) by open surgery
  Interventions: Procedure: open ureteral reimplantation (Lich-Gregoir)

INTERVENTIONS:
Procedure: subureteral endoscopic Injection of Dextranomer/Hyaluronic acid (Dexell) — The subureteral endoscopic injection was done under general anesthesia. the investigators used the subureteral injection technique (STING), as described by O'Donnell and Puri. The volume of Dexell was injected until ureteral orifice collapse in all patients. The needle was held for 30 s.
  Other Names: Dexell subureteral injection
  Arms: Subureteral endoscopic injection
Procedure: open ureteral reimplantation (Lich-Gregoir) — The juxtavesical ureter is dissected by open surgery and a submucosal groove is created extending laterally from the ureteral hiatus along the course of the ureter. The ureter is placed in the groove and the detrusor is closed over the ureter with ureteric stent fixation for 21 days. the surgical wound is closed in layers. Urethral catheter for bladder drainage for 3-5 days.
  Other Names: extra-vesical (Lich-Gregoir) ureteroneocystostomy
  Arms: open ureteral reimplantation (lich-gregoir)

SUMMARY:
In this study, the investigators aim to compare the outcomes of Dextranomer/hyaluronic acid (Dexell®) and extravesical reimplantation (Lich- Gregoir) procedures for primary vesicoureteral reflux (VUR) grades III and IV in children.

DETAILED DESCRIPTION:
A total of 60 patients with 93 renal unites were prospectively enrolled in a comparative intervention study. Patients were randomly allocated by simple randomization at a 1: 1 ratio into 2 groups, where dextranomer/hyaluronic acid (Dexell) injection was used in Group A (30 patients with 45 renal units) and Lich-Gregoir in Group B (30 patients with 48 renal units).

Children over 1 year with primary VUR grade III & IV based on recent VCUG included in the study.

This study and method of attaining consent were approved by clinical research and ethical committee of our department. Written consents were taken from patients' guardians involved in the study. the investigators offered all of patients with symptomatic VUR entry into a prospective protocol between June 2015 and February 2018 at the Urology Department, Al Hussein University Hospital, Al-Azhar University.

Surgical Technique:

1. dextranomer/hyaluronic acid injection: The endoscopic procedure was done under general anesthesia, and all patients received antibiotic prophylaxis. the investigators used the subureteral injection technique (STING), as described by O'Donnell and Puri . The volume of dextranomer/hyaluronic acid was injected until ureteral orifice collapse in all patients. The needle was held for 30 s.
2. ureteral reimplantation (lich-gregoir): The juxtavesical ureter is dissected and a submucosal groove is created extending laterally from the ureteral hiatus along the course of the ureter. The ureter is placed in the groove and the detrusor is closed over the ureter with ureteric stent fixation for 21 days. Urethral catheter for bladder drainage for 3-5 days.

Postoperative Care All children were maintained on prophylaxis until resolution of reflux documented on the VCUG. Patients were assessed by general examination, serial urinalysis and urine C.S. renal ultrasound at 1,3 months and at 1 year after the procedure and a VCUG at 3-6 months. MRU at 1 year. DMSA scintigraphy were done at 6 months after the procedure. the investigators analyzed the outcome in these 2 surgical groups in terms of success rate at short-term follow-up, contralateral reflux, de novo hydronephrosis, urinary tract infections and complications.

The investigators considered that a patient was cured from reflux when there was no VUR on VCUG.

ELIGIBILITY:
Inclusion Criteria:

• Children over one year with primary Vesico-Ureteral reflux grade III and IV.

Exclusion Criteria:

* Secondary Vesico-Ureteral reflux.
* Active urinary tract infection
* Untreated voiding dysfunction.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
surgical success | 2 years
  The outcomes between both groups were analyzed according to surgical success rate. The child was considered to have been cured when there was no reflux on VCUG.

SECONDARY OUTCOMES:
complications | 2 years
  contralateral reflux, de novo hydronephrosis, urinary tract infections and other complications.
median costs | 2 years
  median costs in US dollars compared between two groups

CONTACTS AND LOCATIONS:
Overall Officials: hussein galal, MD, Study Director — professor of urology- department of urology- Al-Azhar faculty of medicine

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in the publication including the Study Protocol Statistical Analysis Plan, Clinical Study Report, and Analytic Code.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: the data will be available 6 months after publication.
Access Criteria: the data will be shared with researchers who provide a methodologically sound proposal to achieve aims in approved proposal. the mechanism of data availability include directing the approved proposal to (elsayedsalih@azhar.edu.eg) also data will be available at our university's warehouse after publication.
URL: http://drive.google.com/drive/u/0/folders/1UiUtebWQHukhJsg6DPXdz0srJHupl43k

REFERENCES:
- [Result] Garcia-Aparicio L, Rovira J, Blazquez-Gomez E, Garcia-Garcia L, Gimenez-Llort A, Rodo J, Morales L. Randomized clinical trial comparing endoscopic treatment with dextranomer hyaluronic acid copolymer and Cohen's ureteral reimplantation for vesicoureteral reflux: long-term results. J Pediatr Urol. 2013 Aug;9(4):483-7. doi: 10.1016/j.jpurol.2013.03.003. Epub 2013 Apr 18. PMID 23602843
- [Result] Karakus SC, User IR, Kilic BD, Akcaer V, Ceylan H, Ozokutan BH. The comparison of dextranomer/hyaluronic acid and polyacrylate-polyalcohol copolymers in endoscopic treatment of vesicoureteral reflux. J Pediatr Surg. 2016 Sep;51(9):1496-500. doi: 10.1016/j.jpedsurg.2016.02.092. Epub 2016 Mar 12. PMID 27061353
- [Derived] Salih EM, Eldamanhory H, Selmy GI, Galal HA. Comparison of Subureteral Endoscopic Injection of Dextranomer/Hyaluronic Acid and Lich-Gregoir Ureteral Reimplantation in the Treatment of Pediatric Primary Vesicoureteral Reflux: A Prospective Randomized Study. J Laparoendosc Adv Surg Tech A. 2021 Jun;31(6):719-723. doi: 10.1089/lap.2020.0973. Epub 2021 Mar 22. PMID 33751917